CLINICAL TRIAL: NCT03705767
Title: The Maternal-fetal Gradient of Free and Esterified Phytosterols in Term Human Pregnancy at Delivery
Brief Title: Placental Passage of Free and Esterified Phytosterols in Humans
Acronym: PTS
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Virgilio Paolo Carnielli, MD, Phd, Professor of Neonatal Pediatrics, Università Politecnica delle Marche
Other Study IDs: PTS1
Record Dates: First submitted 2017-11-13; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Mother Fetus Relations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Total plasma cholesterol rises by 60 % with progressing pregnancy in humans. Because lipid-lowering drugs are contraindicated during pregnancy, natural compounds, such as phytosterols, may be a safe and effective alternative to prevent undesirable effects. Information on phytosterols in pregnancy is so far very limited. To date, to the best of our knowledge, no studies have characterized the maternal-fetal gradient of free and esterified phytosterols in full-term human pregnancy. For this purpose, maternal and cord blood cholesterol and non-cholesterol sterol (campesterol, stigmasterol, sitosterol) concentrations were measured in term pregnant women at delivery by using gas chromatography-mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* A single pregnancy
* A gestational age determined from known last maternal menstrual period higher than 37 weeks
* A normal diet without phytosterol supplementation during pregnancy
* Written informed consent available.

Exclusion Criteria:

* Major congenital anomalies
* Maternal history of cardiovascular disease
* Endocrine disorders such as diabetes, hypercholesterolemia, pre-eclampsia, thyroid or adrenal problems
* Clinical chorioamnionitis

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Free and esterified phytosterol ratio | the day of delivery
  Plasma free and esterified phytosterol concentrations will be measured in mother-cord blood pairs at delivery. Plasma phytosterol concentrations will be the sum of plasma campesterol, stigmasterol and sitosterol concentrations (mg/L). Gas chromatography-mass spectrometry will be used for measurements.

SECONDARY OUTCOMES:
total cholesterol concentrations | the day of delivery
  plasma cholesterol concentrations (mg/L) will be measured to evaluate the cholesterol metabolism in mother-cord blood pairs at delivery. Total cholesterol in pregnant women and cord blood will be calculated from plasma free and esterified cholesterol. Cholesterol concentrations will be measured by using gas chromatography-mass spectrometry.
total lathosterol concentrations | the day of delivery
  plasma lathosterol concentrations (mg/L) will be measured to evaluate the cholesterol metabolism in mother-cord blood pairs at delivery. Total lathosterol in pregnant women and cord blood will be calculated from plasma free and esterified lathosterol. Lathosterol concentrations will be measured by using gas chromatography-mass spectrometry.
total 7-dehydrocholesterol concentrations | the day of delivery
  plasma 7-dehydrocholesterol concentrations (mg/L) will be measured to evaluate the cholesterol metabolism in mother-cord blood pairs at delivery. Total 7-dehydrocholesterol in pregnant women and cord blood will be calculated from plasma free and esterified 7-dehydrocholesterol.
  7-dehydrocholesterol concentrations will be measured by using gas chromatography-mass spectrometry.
total 7-alpha-hydroxycholesterol concentrations | the day of delivery
  plasma 7-alpha-hydroxycholesterol concentrations (mg/L) will be measured to evaluate the cholesterol metabolism in mother-cord blood pairs at delivery. Total 7-alpha-hydroxycholesterol in pregnant women and cord blood will be calculated from plasma free and esterified 7-alpha-hydroxycholesterol. 7-alpha-hydroxycholesterol concentrations will be measured by using gas chromatography-mass spectrometry.
fatty acid concentrations | the day of delivery
  plasma fatty acid concentrations (mg/dl) will be measured to evaluate the fat metabolism in mother-cord blood pairs at delivery. Total fatty acids will be measured by using gas chromatography with flame ionization detector will be used for the measurement of fatty acids.

REFERENCES:
- [Background] Montelongo A, Lasuncion MA, Pallardo LF, Herrera E. Longitudinal study of plasma lipoproteins and hormones during pregnancy in normal and diabetic women. Diabetes. 1992 Dec;41(12):1651-9. doi: 10.2337/diab.41.12.1651. PMID 1446807
- [Background] Rideout TC, Movsesian C, Tsai YT, Iqbal A, Raslawsky A, Patel MS. Maternal Phytosterol Supplementation during Pregnancy and Lactation Modulates Lipid and Lipoprotein Response in Offspring of apoE-Deficient Mice. J Nutr. 2015 Aug;145(8):1728-34. doi: 10.3945/jn.115.215061. Epub 2015 Jun 17. PMID 26084365
- [Background] Berger A, Jones PJ, Abumweis SS. Plant sterols: factors affecting their efficacy and safety as functional food ingredients. Lipids Health Dis. 2004 Apr 7;3:5. doi: 10.1186/1476-511X-3-5. PMID 15070410
- [Background] Piccoli GB, Clari R, Vigotti FN, Leone F, Attini R, Cabiddu G, Mauro G, Castelluccia N, Colombi N, Capizzi I, Pani A, Todros T, Avagnina P. Vegan-vegetarian diets in pregnancy: danger or panacea? A systematic narrative review. BJOG. 2015 Apr;122(5):623-33. doi: 10.1111/1471-0528.13280. Epub 2015 Jan 20. PMID 25600902
- [Background] Gao F, Wang G, Wang L, Guo N. Phytosterol nutritional supplement improves pregnancy and neonatal complications of gestational diabetes mellitus in a double-blind and placebo-controlled clinical study. Food Funct. 2017 Jan 25;8(1):424-428. doi: 10.1039/c6fo01777k. PMID 28091647
- [Result] Nikkila K, Riikonen S, Lindfors M, Miettinen TA. Serum squalene and noncholesterol sterols before and after delivery in normal and cholestatic pregnancy. J Lipid Res. 1996 Dec;37(12):2687-95. PMID 9017519
- [Result] Miettinen HE, Rono K, Koivusalo S, Stach-Lempinen B, Poyhonen-Alho M, Eriksson JG, Hiltunen TP, Gylling H. Elevated serum squalene and cholesterol synthesis markers in pregnant obese women with gestational diabetes mellitus. J Lipid Res. 2014 Dec;55(12):2644-54. doi: 10.1194/jlr.P049510. Epub 2014 Oct 9. PMID 25301963
- [Result] Vuorio AF, Miettinen TA, Turtola H, Oksanen H, Gylling H. Cholesterol metabolism in normal and heterozygous familial hypercholesterolemic newborns. J Lab Clin Med. 2002 Jul;140(1):35-42. doi: 10.1067/mlc.2002.125214. PMID 12080326